CLINICAL TRIAL: NCT03043885
Title: Ridge Preservation With Platelet Rich Fibrin Augmented With Freeze Dried Bone Allograft: A Comparative Clinical, Histological, and Micro-computed Tomography Study
Brief Title: Ridge Preservation With Platelet Rich Fibrin Augmented With Freeze Dried Bone Allograft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Mark Ryder, Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-13360
Record Dates: First submitted 2017-02-01; First posted 2017-02-06 (Estimated); Results first posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Alveolar Ridge Preservation
MeSH Terms: interventions — Blood Coagulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- PRF (Experimental)
  Interventions: Device: PRF
- PRF+FDBA (Experimental)
  Interventions: Device: FDBA; Device: PRF
- FDBA (Active Comparator)
  Interventions: Device: FDBA
- Blood Clot (Active Comparator)
  Interventions: Procedure: Blood Clot

INTERVENTIONS:
Device: FDBA — Graft material used to graft extraction socket
  Arms: FDBA; PRF+FDBA
Device: PRF — Autologous blood product used to graft extraction socket
  Arms: PRF; PRF+FDBA
Procedure: Blood Clot — Surgical treatment of extraction socket without addition of graft material
  Arms: Blood Clot

SUMMARY:
Improved predictability and quality of bone healing after a tooth is removed is clinically relevant, in that, it improves our ability to achieve successful implant placement at edentulous sites. Currently, a variety of grafting materials and biologic agents are utilized clinically to improve bone healing and provide sufficient dimensions of bone to support a dental implant. Platelet rich fibrin (PRF) is one such product that can be used for this application. PRF is a concentrated blood product attained from the patient's own blood consisting of a natural bioscaffold with integrated growth factors capable of sustained release. Once processed, PRF is implanted back into the patient at the wound or defect site to encourage healing. The literature regarding PRF is currently dominated by heterogeneous applications of PRF for reparative and regenerative therapies without a consensus of its clinical efficacy and appropriate application. In this clinical study, PRF will be evaluated to ascertain its clinical efficacy in improving bone formation and alveolar dimensional stability after tooth extraction. A classic bone grafting material used for this purpose, freeze dried bone allograft (FDBA), will be incorporated with the PRF or compared directly to PRF alone. It is hypothesized that the natural scaffold and incorporated growth factors of PRF augmented with the solubility resistance of FDBA will function as an ideal bioscaffold to promote bone healing to a greater extent compared to PRF, FDBA, or blood clot alone.

DETAILED DESCRIPTION:
This is a randomized controlled clinical study evaluating the efficacy of four treatment modalities for ridge preservation after extraction of a tooth in preparation for dental implant placement. After tooth extraction the alveolar crest remodels during healing with reductions in vertical and horizontal dimensions. The resulting reduced dimensions after healing of the alveolar crest may be inadequate to successfully place a dental implant to replace the missing tooth. In an attempt to minimize the reductions in dimensions and provide mature healthy bone to support the dental implant, different ridge preservation techniques (treatment of the extraction socket) have been utilized.

Forty subject from the UCSF Dental School who will be having a tooth extracted and replaced with a dental implant will be randomly assigned into the four ridge preservation treatment groups. After three months of healing bone samples from the ridge preservation site will be collected during the implant placement when bone is removed during the osteotomy preparation for the implant. Samples will be evaluated for the extent and quality of bone healing via histomorphometric and micro-CT analysis. Clinical measures of alveolar ridge dimensions will be taken before and after tooth extraction to determine extent of dimensional stability under the different treatment groups.

The four treatments modalities for ridge preservation include autologous platelet rich fibrin (PRF), PRF+freeze dried bone allograft (FDBA), FDBA, collagen barrier membrane. Subjects will be enrolled in the study from the time the socket treated to the time of implant placement (3 months). The results of this study will help to elucidate the extent and quality of bone healing using four different methods for ridge preservation in preparation for implant placement. Further, this study will advance our knowledge of PRF, an autologous sourced blood product used in dentoalveolar surgeries with proven in-vitro qualities but still requiring more extensive clinical testing to demonstrate its full clinical utility.

ELIGIBILITY:
Inclusion Criteria:

1. Single rooted teeth requiring extraction
2. Intact buccal and lingual plate within approximately 3-4 mm from gingival crest
3. No clinical or radiographic signs of periapical pathology
4. Acceptable oral hygiene

Exclusion Criteria:

1. Unable to comply with necessary scheduled visits
2. Poor oral hygiene
3. Failing/failed endodontic treatment with history/presence of sinus tracts
4. Pregnant woman or patients who intend to become pregnant
5. Tobacco use
6. Immunosuppressed
7. Type I or type II diabetes
8. Patient with any blood disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01-05 (Actual); Primary Completion 2016-05-09 (Actual); Study Completion 2017-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ryder, DDS, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Platelet-rich Fibrin: PRF: Autologous blood product used to graft extraction socket
Period: Overall Study
Arm/Group | Platelet-rich Fibrin | PRF+FDBA | FDBA | Blood Clot
Started | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Platelet-rich Fibrin | PRF+FDBA | FDBA | Blood Clot | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 8 | 8 | 29
  >=65 years | 3 | 4 | 2 | 2 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 5 | 5 | 22
  Male | 4 | 4 | 5 | 5 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 10 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Vital Bone
Description: Percentage of vital bone at healed extraction socket
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of vital bone
Arm/Group | Platelet-rich Fibrin | PRF+FDBA | FDBA | Blood Clot
Number analyzed (Participants) | 10 | 10 | 10 | 10
percentage of vital bone | 46 (18) | 39 (10) | 29 (14) | 40 (15)

2. Secondary Outcome: Bone Mineral Density
Description: The bone mineral density (measured via micro-CT) at healed extraction sockets
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mg/cm3
Arm/Group | Platelet-rich Fibrin | PRF+FDBA | FDBA | Blood Clot
Number analyzed (Participants) | 10 | 10 | 10 | 10
mg/cm3 | 493 (70) | 521 (58) | 487 (64) | 551 (58)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Platelet-rich Fibrin | PRF+FDBA | FDBA | Blood Clot
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No